CLINICAL TRIAL: NCT04787393
Title: Lancashire Objective Volume Evaluation of Leg Oedema in Heart Failure Second (LOVE-HF-2)
Brief Title: Lancashire Objective Volume Evaluation of Leg Oedema in Heart Failure Second Pilot
Acronym: LOVE-HF-2
Status: Completed | Type: Observational
Sponsor: Heartfelt Technologies (Industry)
Collaborators: Blackpool Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: BTH01.2
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Edema leg; Quality of life; Hospital Admissions; Days alive out of hospital; Heartfelt Device; Artificial Intelligence
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LOVE-HF-2 Participants: Participants will have the Heartfelt device as well as a set of weighing scales installed at home.
  Alerts will be raised for the patient to be seen at home or in clinic by clinician ( the clinician will be blinded to the type of alert). During this face-to-face encounter, the clinician will perform a detailed oedema assessment (recording pitting depth, time of recovery, height oedema, overall grading), ankle circumference measurement, weight measurements, and echo (Left ventricular ejection fraction, Left atrial volumes, inferior vena cava diameter, Diastolic function (E/A, E/E'), TAPSE and TR jet velocity + visually estimated mitral and tricuspid regurgitation).
  Interventions: Device: Heartfelt device; Device: Connected weighing scales

INTERVENTIONS:
Device: Heartfelt device — The Heartfelt device uses a system of scanner in a compact device to generate depth images of the feet and lower legs with a view to detecting early volume changes. The device can be installed on the wall or as a free standing unit, For the measurements to take place, the participant walks in the field of view of the device, measurments are only taken when the patients has bare feet and no slippers/shoes, so the location of the device in the home is choosen to match this requirement. Participants are not expected to change anything to their routine. The device can also take measurements in the dark.
Device: Connected weighing scales — The participant will be instructed to use those scales for the period of the study, as often as directed by their healthcare professional. The weighing scales display weight so that the participants can record the weight in their own heart failure records if they wish to do so.
  The scales will communicate with the Personal Computer (PC) contained in the Heartfelt device and the data will be sent to the Heartfelt server through an encrypted link.
  The data from the scales will be reviewed retrospectively, as the comparison in this study is with standard care, not with enhanced provision of care, which would be the case if we were using automatic reporting of weights.

SUMMARY:
Patients with heart failure (HF) who recently received treatment with IV diuretics for worsening congestion or outpatients with HF and peripheral oedema treated with at least 80 mg furosemide (or equivalent)/day will be recruited in the LOVE-HF-2 trial at Blackpool Victoria Hospital. The main objective of the study is to test if the Heartfelt device is sensitive to change across the full range of the individual patient's oedema. The participants will be given the Heartfelt device to use in their home. This device automatically and passively measures patient's foot and lower leg's volume without the patient having to remember to do anything. The patients will be seen face to face with a cardiologist to evaluate peripheral oedema using standard clincial technics as well as overall congestion level. The investigators aim to recruit 30 participants for the observational pilot study.

The study follows its sister pilot trial, LOVE-HF (NCT04787380).

DETAILED DESCRIPTION:
Heart Failure is the final common pathway of most forms of cardiovascular disease. In the United Kingdom (UK), it affects around 900 000 people, causes or complicates around 5% of adult emergency hospital admissions and consumes up to 2% of total National Health Service (NHS) expenditure. An important part of discharge planning includes measures such as early follow up in order to prevent readmissions. The hallmark of heart failure is fluid retention and between 2009 and 2016, 43% to 50% of hospital admissions were associated with peripheral oedema. Therefore, early recognition of this and treatment of the congestion may prevent hospital admissions. In clinical trials, management strategies have included patient education, telemedicine and remote monitoring. The main non-invasive method for detecting fluid retention has been the use of weight as a surrogate marker.

The Heartfelt device is an invention that uses a system of cameras in a compact device in order to generate 3 dimensional images of the feet and lower legs. The volumes can then be calculated and thus, changes in amount of peripheral oedema can be estimated. In a clinical trial (NCT02993601) performed by the Heart Failure team at the Royal Brompton Hospital, there was good correlation between measurements made by Heartfelt and a water displacement method. The resolution was as good as 20mls.

By positioning the Heartfelt device in the bedroom, automatic measurements can be made whenever the subject gets in and out of bed. Images are only taken of the specified subject. Data is censored so that the part of the body which is 50cm above the floor is not stored. Encrypted, anonymised data is transmitted over the internet to the company's secure servers. Personal identifiable data (participant name, address, age…) is stored on an encrypted hard drive, along with linkage information (device serial numbers) to associate the participant identifiable data with the data captured in the home. Therefore, data collection is not only secure but entirely passive, which is a major advantage compared with previous non-invasive methods and it is applicable to a very wide range of compliant and non-compliant patients.

The LOVE-HF trial (NCT04787380) demonstrated that the number of days with missing data collected by the Heartfelt device was significantly lower than that of the weighing scales, providing a promising tool for home patient monitoring.

Being able to demonstrate that the device can provide a measure of oedema that is clinically relevant over the full range of individual patient's oedema is the main objective of this study as this will further adds to the validation of the device.

ELIGIBILITY:
Inclusion criteria:

Patients with HF who recently (< 6 months) received treatment with IV diuretics for worsening congestion or outpatients with HF and peripheral oedema (any degree) who are treated with at least 80 mg furosemide (or equivalent) orally per day Patients with HF older than 18 years Patients who took part in LOVE-HF can also be approached.

The research team will try to include as many patients as possible in the month following discharge, however we will not exclude consideration of a small proportion of patients within 6 months of decompensation. This has the extra advantage of demonstrating the value of the device beyond 1-2 months of decompensation.

Exclusion Criteria:

1. Inability to provide informed consent*
2. Participant has bandages to lower limbs everyday
3. Participant has an amputation of the foot
4. Participant is a regular wheelchair user
5. Participant is of no fixed abode
6. Participant has a potentially reversible cause of decompensated heart failure and is awaiting urgent intervention (revascularisation/ valvular heart disease), which means the patient cannot be discharged for home-based care
7. Participant is taking part in a conflicting evaluation/study that could confound the results of this evaluation and/or impact clinical interventions and participant outcomes
8. Participant must not be pregnant, and is taking relevant birth control if of child-bearing potential*

Note that a participant not able to comply with weighing, or questionnaires is NOT an exclusion criteria as the Heartfelt device should provide data for these participants despite their lack of ability to adhere to the usual monitoring protocol, and this is seen as one of the long term benefits that the device can provide.

* This exclusion criteria (a) has been added as participants would need to be able to communicate directly with the Heartfelt team, etc.
* This exclusion criteria (h) has been requested by the insurance provider for clinical trial cover.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be chosen to be close representatives of the target population for the device: Heart failure patients at high risk of decompensation, with associated peripheral oedema.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Foot volume measured by the Heartfelt device in the home. | 1-6 months
Foot volume measured by the Heartfelt device in the hospital. | 1-6 months

SECONDARY OUTCOMES:
Patient weight measured in hospital. | 1-6months
Oedema/Edema scores | 1-6months
  The clinical oedema scores is a matrix of oedema eight, depth at each of the prespecified location on the leg and time for recovery at each of the prespecified (Brodovicz et al., Clin Med Res 2009). The time for recovery is presented in seconds for each prespecified location on each leg. The depth is presented in millimeters for each prespecified location on each leg.
  The NICOR oedema score (No, Mild, Moderate, Severe) is also recorded. A bespoke scale is also used to record oedema height (0=None, 1=Includes ankle but non higher; 2=Above ankle, up to and including the knee; 3=Above the knee)
Left ventricular ejection fraction | 1-6months
Left atrial volume | 1-6months
Diastolic function (E/A, E/E') | 1-6months
Inferior vena cava diameter | 1-6months
TAPSE and TR jet velocity | 1-6months
visually estimated mitral and tricuspid regurgitation | 1-6months
Ankle circumference | 1-6months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cassidy, Principal Investigator — Blackpool Teaching Hospitals NHS Foundation Trust
Locations (1):
- Department of Cardiology, Lancashire Cardiac Centre, Blackpool Teaching Hospital, Blackpool, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No